CLINICAL TRIAL: NCT03904979
Title: Writing to Reduce Stress in Expectant Moms: The RESet Study
Brief Title: Therapeutic Writing to Reduce Stress
Acronym: RESeT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to continue due to loss of staff.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-2187
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Complications; Stress, Physiological; High Risk Pregnancy
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Participants will have identical journals regardless of the intervention or control group status, and providers will be blinded to the writing prompts that participants are given. Women who are randomized to 'no writing' will be provided a blank journal without any instruction. this will be considered a 'gift' for study participation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic Writing Prompts (Experimental): Participants will be given writing prompts that discuss events that have been perceived as stressful in their lives and how they may or may not have cultivated resilience and coping strategies because of it.
  Interventions: Other: Writing exercises
- General Writing Prompts (Placebo Comparator): Participants will be given writing prompts that discuss "neutral" topics unrelated to their life stress, resilience, or coping.
  Interventions: Other: Writing exercises
- No Writing (No Intervention): Participants will not be given writing prompts during their prenatal care. They will be given blank journals that will NOT contain any instructions or writing prompts.

INTERVENTIONS:
Other: Writing exercises — Participants will be given journals with writing prompts to be completed throughout their pregnancy.
  Arms: General Writing Prompts; Therapeutic Writing Prompts

SUMMARY:
Purpose: The investigators hypothesize that exposure to chronic environmental stress is a risk factor for adverse pregnancy outcomes related to preterm birth and preeclampsia among high-risk pregnant women. Additionally, the investigators hypothesize that women can be screened for high levels of environmental stress through the perceived stress scale, and therapeutic writing can be used as a low-resource intervention to help decrease maternal perceived stress and inflammation - measured through analysis of maternal serum and placental samples.

Participants: Pregnant women at high risk for adverse pregnancy outcomes, including pre-eclampsia and preterm birth, enrolled in prenatal care at UNC will be recruited for participation

Procedures: Using results from the perceived stress scale, the investigators will identify women who screen positive for high environmental stress. Women meeting inclusion criteria will be contacted for possible participation at regularly scheduled prenatal visits. Women who are enrolled will be randomized to generalized writing prompts, therapeutic writing prompts, or no writing during their pregnancy to be administered at each prenatal visit. Maternal blood sample for biochemical markers of stress and gene expression will be obtained at the initial visit; a followup blood sample will be obtained later in pregnancy, and a small portion of the placenta saved at delivery. Delivery outcomes will be obtained through medical record review.

DETAILED DESCRIPTION:
During pregnancy, women regularly interact with healthcare professionals, an often untapped resource and opportune time to optimize mental health, positively impacting outcomes. Cumulative psychosocial stress is a risk factor for several adverse obstetric outcomes including preterm birth (PTB), preeclampsia, fetal growth restriction, and postpartum depression.

The overarching hypothesis of this study is that pregnant women with high levels of stress can be identified through easily-implemented screening tools; importantly, the investigators propose that these women can be engaged in care via a cost-effective therapeutic writing intervention combined with the availability of expert pastoral and perinatal psychiatry resources.

Women will be enrolled early in pregnancy and followed prospectively. Some women (if randomized to a writing group) will complete a standardized writing prompt at several time points during gestation. The investigators will follow their outcomes prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Women will be prospectively recruited.

  1. Gestational age: All women presenting for prenatal care at 8.0 to 19.9 weeks' gestation through the UNC-Hospitals High Risk obstetrics clinic will be screened for high risk of an adverse pregnancy outcome (ex: preterm birth or pre-eclampsia) through review of their medical record.
  2. Singleton viable intrauterine pregnancy, with dating confirmed by ultrasound or plans for ultrasound to confirm dating prior to study enrollment
  3. No structural abnormalities or aneuploidy
  4. Ability to communicate in and provide consent in English
  5. Women with at least ONE of the following high risk criteria:

     a. Short cervix by endovaginal ultrasound, measuring <25mm b. Prior spontaneous preterm birth 16.0 - 33.9 weeks' gestation i. Documentation of the prior spontaneous preterm birth in the patient's medical records is desirable but is not required for eligibility.

     ii. The previous preterm delivery cannot be an antepartum stillbirth but an intrapartum stillbirth (due to extreme prematurity) is allowable.

     c. Chronic hypertension on medications d. History of pre-eclampsia requiring delivery <37 weeks' gestation, or history of severe pre-eclampsia delivering at any gestational age

     OR
  6. Women with at least TWO of the following moderate risk criteria:

     1. Prior preterm birth 34.0-36.9 weeks
     2. Chronic hypertension not requiring medications
     3. History of term pre-eclampsia
     4. Type II diabetes on insulin
     5. Obesity with a BMI >30
     6. Smoking during pregnancy
     7. Black race
     8. Maternal age <18 years old or >40 years old
     9. Nulliparous
     10. Uninsured, or medicaid insurance
  7. Women who meet at least one major or 2 minor inclusion criteria along with the other criteria above will then be screened for high levels of acute and chronic stress and trauma using the Perceived Stress questionnaire to determine final eligibility for the study

Exclusion Criteria:

1. Persistent Illicit drug or alcohol abuse during current pregnancy >12 weeks. Use of tobacco and/or marijuana is not an exclusion. Methadone or suboxone use in an approved treatment program is not an exclusion.
2. Prior preterm birth or preeclampsia was in a pregnancy complicated by fetal aneuploidy or major congenital fetal anomalies in the absence of another pregnancy meeting above inclusion criteria
3. Major congenital anomaly such as major structural deficit of the heart, lungs, or brain or aneuploidy

   1. Mild renal abnormalities, clubfoot, isolated cleft lip/palate, etc. in the fetus are not a reason for exclusion
   2. For a detailed list of major anomalies, see Table 3 - Major Fetal Anomalies / Congenital Malformations, below. Two or more minor anomalies observed together (see Table 2 - Minor Fetal Anomalies / Congenital Malformations) count as a "major" anomaly
   3. Isolated 'soft markers' for aneuploidy (such as choroid plexus cysts, echogenic bowel, etc.) are not a reason for exclusion
   4. If aneuploidy screening is performed, any aneuploidy screen positive test with a risk for aneuploidy greater than 1 in 25 without negative confirmatory definitive aneuploidy testing is reason for exclusion
4. Spanish speaking women
5. Women participating in other intervention-based studies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Percent Participation in Writing Activity | through study completion, an average of 7 months per participant and 2 years for entire study
  The percentage of women who respond that they completed their assigned writing activity will be measured.
Statistically significant improvement (reduction) in the Perceived Stress Scale Score | through study completion, an average of 7 months per participant and 2 years for entire study
  Psychological instrument used to measure one's perception of stress (score range 0-40) will be assessed before and after the assigned writing activity. Higher scores on the scale indicate a higher vulnerability for those with a high levels of perceived stress in their life. Prior studies have noted the average score for a female age 30-44 is approximately 14.
Proportion of women with adverse perinatal outcomes | outcome will be ascertained at delivery
  We will define adverse pregnancy outcomes as a composite of preterm birth <37 weeks, intrauterine growth restriction, preeclampsia, and placental abruption; outcomes will be compared between randomization groups
Change in pro-inflammatory biomarkers in maternal blood by randomization group | through study completion, an average of 7 months per participant and 2 years for entire study
  All women participating in the study will have a blood draw. Levels of stress biomarkers (e.g., interleukin-6) will be compared by randomization group
Change in pro-inflammatory biomarkers in maternal blood by outcome | through study completion, an average of 7 months per participant and 2 years for entire study
  All women participating in the study will have a blood draw. Levels of stress biomarkers (e.g., interleukin-6) will be compared between women who develop the adverse perinatal outcome and those who do not
Change in stress-related gene expression in maternal blood by randomization group | through study completion, an average of 7 months per participant and 2 years for entire study
  All women participating in the study will have a blood draw. We will evaluate gene expression of the CTRA gene panel (conserved transcriptional response to adversity gene panel) by randomization group
Change in stress-related gene expression in maternal blood by outcome | through study completion, an average of 7 months per participant and 2 years for entire study
  All women participating in the study will have a blood draw. We will evaluate gene expression of the CTRA gene panel (conserved transcriptional response to adversity gene panel) by whether or not the patient developed the adverse perinatal outcome

SECONDARY OUTCOMES:
Utilization of professional psychiatric care | through study completion, an average of 7 months per participant and 2 years for entire study
  proportion of women who initiate or continue therapy with professional psychiatric care provider
Stress related pathways gene expression - placental tissue - by randomization group | through study completion, an average of 7 months per participant and 2 years for entire study
  After delivery, we will evaluate whether there are differences in the conserved transcriptional response to adversity gene panel (CTRA gene panel) by randomization groups
Stress related pathways gene expression - placental tissue - by diagnosis of adverse perinatal outcome | through study completion, an average of 7 months per participant and 2 years for entire study
  After delivery, we will evaluate whether there are differences in the conserved transcriptional response to adversity gene panel (CTRA gene panel) by whether or not the patient developed the adverse perinatal outcome
Rate of preterm birth less than 37 weeks' gestation by randomization group | through study completion, an average of 7 months per participant and 2 years for entire study
  we will individually evaluate the outcomes of preterm birth <37 weeks, intrauterine growth restriction, preeclampsia, and placental abruption; outcomes will be compared between randomization groups
Rate of diagnosis of intrauterine growth restriction, using sex-specific curves, by randomization group | through study completion, an average of 7 months per participant and 2 years for entire study
  we will individually evaluate the outcomes of preterm birth <37 weeks, intrauterine growth restriction, preeclampsia, and placental abruption; outcomes will be compared between randomization groups
Rate of diagnosis of preeclampsia by randomization group | through study completion, an average of 7 months per participant and 2 years for entire study
  we will individually evaluate the outcomes of preterm birth <37 weeks, intrauterine growth restriction, preeclampsia, and placental abruption; outcomes will be compared between randomization groups
Rate of diagnosis of placental abruption by randomization group | through study completion, an average of 7 months per participant and 2 years for entire study
  we will individually evaluate the outcomes of preterm birth <37 weeks, intrauterine growth restriction, preeclampsia, and placental abruption; outcomes will be compared between randomization groups

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A Manuck, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Women's Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
All information that is collected for this study will be stored in locked filing cabinets and/or offices and on the secure UNC server on the RedCap database. Participants will be assigned a unique study-id number for this study. Only the PI and Sponsor for the study will have access to the key linking this study id number to their personal clinical information and identifiers.

REFERENCES:
- [Background] McEwen BS. Stress, adaptation, and disease. Allostasis and allostatic load. Ann N Y Acad Sci. 1998 May 1;840:33-44. doi: 10.1111/j.1749-6632.1998.tb09546.x. PMID 9629234
- [Background] Geronimus AT, Hicken M, Keene D, Bound J. "Weathering" and age patterns of allostatic load scores among blacks and whites in the United States. Am J Public Health. 2006 May;96(5):826-33. doi: 10.2105/AJPH.2004.060749. Epub 2005 Dec 27. PMID 16380565
- [Background] Schulkin J, Gold PW, McEwen BS. Induction of corticotropin-releasing hormone gene expression by glucocorticoids: implication for understanding the states of fear and anxiety and allostatic load. Psychoneuroendocrinology. 1998 Apr;23(3):219-43. doi: 10.1016/s0306-4530(97)00099-1. PMID 9695128
- [Background] Anding JE, Rohrle B, Grieshop M, Schucking B, Christiansen H. Couple comorbidity and correlates of postnatal depressive symptoms in mothers and fathers in the first two weeks following delivery. J Affect Disord. 2016 Jan 15;190:300-309. doi: 10.1016/j.jad.2015.10.033. Epub 2015 Oct 28. PMID 26546770
- [Background] Edwards B, Galletly C, Semmler-Booth T, Dekker G. Does antenatal screening for psychosocial risk factors predict postnatal depression? A follow-up study of 154 women in Adelaide, South Australia. Aust N Z J Psychiatry. 2008 Jan;42(1):51-5. doi: 10.1080/00048670701739629. PMID 18058444
- [Background] Juul SH, Hendrix C, Robinson B, Stowe ZN, Newport DJ, Brennan PA, Johnson KC. Maternal early-life trauma and affective parenting style: the mediating role of HPA-axis function. Arch Womens Ment Health. 2016 Feb;19(1):17-23. doi: 10.1007/s00737-015-0528-x. Epub 2015 May 9. PMID 25956587
- [Background] Meltzer-Brody S, Boschloo L, Jones I, Sullivan PF, Penninx BW. The EPDS-Lifetime: assessment of lifetime prevalence and risk factors for perinatal depression in a large cohort of depressed women. Arch Womens Ment Health. 2013 Dec;16(6):465-73. doi: 10.1007/s00737-013-0372-9. Epub 2013 Aug 1. PMID 23904137
- [Background] Oh W, Muzik M, McGinnis EW, Hamilton L, Menke RA, Rosenblum KL. Comorbid trajectories of postpartum depression and PTSD among mothers with childhood trauma history: Course, predictors, processes and child adjustment. J Affect Disord. 2016 Aug;200:133-41. doi: 10.1016/j.jad.2016.04.037. Epub 2016 Apr 20. PMID 27131504
- [Background] McDonald SW, Kingston D, Bayrampour H, Dolan SM, Tough SC. Cumulative psychosocial stress, coping resources, and preterm birth. Arch Womens Ment Health. 2014 Dec;17(6):559-68. doi: 10.1007/s00737-014-0436-5. Epub 2014 Jun 20. PMID 24948100
- [Background] Meshberg-Cohen S, Svikis D, McMahon TJ. Expressive writing as a therapeutic process for drug-dependent women. Subst Abus. 2014;35(1):80-8. doi: 10.1080/08897077.2013.805181. PMID 24588298
- [Background] Blasio PD, Camisasca E, Caravita SC, Ionio C, Milani L, Valtolina GG. THE EFFECTS OF EXPRESSIVE WRITING ON POSTPARTUM DEPRESSION AND POSTTRAUMATIC STRESS SYMPTOMS. Psychol Rep. 2015 Dec;117(3):856-82. doi: 10.2466/02.13.PR0.117c29z3. Epub 2015 Nov 23. PMID 26595300
- [Background] Smyth JM, Hockemeyer JR, Tulloch H. Expressive writing and post-traumatic stress disorder: effects on trauma symptoms, mood states, and cortisol reactivity. Br J Health Psychol. 2008 Feb;13(Pt 1):85-93. doi: 10.1348/135910707X250866. PMID 18230238
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629